CLINICAL TRIAL: NCT01565915
Title: Efficacy and Safety of Perlane-L in the Correction of Midface Volume Deficit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medicis Global Service Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA-1400-05
Record Dates: First submitted 2012-03-12; First posted 2012-03-29 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Facial Volume

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Perlane-L (Experimental): Perlane-L treatment
  Interventions: Device: Perlane-L
- Non-Treatment (Sham Comparator): Non-Treatment Arm
  Interventions: Other: Non-treatment

INTERVENTIONS:
Device: Perlane-L — Perlane-L Injection in the midface
  Arms: Perlane-L
Other: Non-treatment — Non-treatment Arm
  Arms: Non-Treatment

SUMMARY:
The purpose of this study is to determine if Perlane-L is safe in increasing cheek volume.

ELIGIBILITY:
Inclusion Criteria:

* Loss of Fullness in Midface Area
* Other items as identified in the protocol

Exclusion Criteria:

* History of allergy or hypersensitivity to injectable hyaluronic acid gel or lidocaine.
* Other items as identified in the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Facial fullness using midface scale | Week 8
  Change in facial fullness using midface scale.

SECONDARY OUTCOMES:
Facial fullness using the midface scale | Up to 12-months post treatment
  Change in facial fullness using midface scale.
Subject satisfaction using the GAIS | Up to 12-months post treatment
  Compare treatment satisfaction as compared to no treatment, on the Global Aesthetic Improvement Scale (GAIS)
Aesthetic improvement | Up to 12-months post treatment
  A subjective assessment of aesthetic improvement post baseline

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Beverly Hills, California
  - San Francisco, California
  - Vista, California
  - Aventura, Florida
  - Coral Gables, Florida
  - Chicago, Illinois
  - Hunt Valley, Maryland
  - Chestnut Hill, Massachusetts
  - Mount Kisco, New York
  - New York, New York
  - Eugene, Oregon